CLINICAL TRIAL: NCT01120002
Title: Efficacy and Safety of Tamibarotene (OAM80) for Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka City University (Other)
Responsible Party: Takami Miki, MD, Professor, Department of Geriatrics and Neurology, Osaka City University Graduate School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OAM80-01
Record Dates: First submitted 2010-04-30; First posted 2010-05-10 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Alzheimer's Disease
Keywords: mild to moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tamibarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo pill (Placebo Comparator)
  Interventions: Drug: Placebo
- Tamibarotene (Active Comparator)
  Interventions: Drug: Tamibarotene

INTERVENTIONS:
Drug: Tamibarotene — Two Tamibarotene 2 mg or placebo tablet per day, once daily.
  Arms: Tamibarotene
Drug: Placebo — Two Tamibarotene 2 mg or placebo tablet per day, once daily.
  Arms: Placebo pill

SUMMARY:
A double blind, placebo-controlled randomized study to evaluate the efficacy and safety of orally administered Tamibarotene to patients of Alzheimer's Disease

DETAILED DESCRIPTION:
Tamibarotene is a synthetic retinoid presently approved in Japan for the treatment of APL, which has a higher receptor selectivity and activity for the Retinoic Acid Receptor subtypes compared to the natural retinoid.

Tamibarotene decreased insoluble amyloid-beta (Ab) 42 deposition in APP mice, and also increased TTR, VAChT and ACh in the brain of SAMP8 mice, which suggest the enhancement of neurotransmission. In the behavioral model such as reduced anxiety of SAMP8 mice and rat passive avoidance test, tamibarotene showed improvement.

Tamibarotene as in other retinoids are known to moderate the immune system and reduce inflammatory cytokines and chemokines, which may control the excessive stimulation of astrocyte and microglia around the Ab plaque. Tamibarotene reduced cytokines and showed clinical efficacy in the rat experimental autoimmune encephalitis model.

Furthermore, retinoids are known to have critical roles during the regeneration stage in the differentiation from neural stem cells (NSC).

In spinal cord injured rats treated with tamibarotene showed better recovery compared to the control.

By these preclinical results, we plan by this study to evaluate the efficacy together with the safety of tamibarotene to the patients of Alzheimer's Disease.

Tamibarotene is used clinically in Japan since 2005. It's side effects are known to be similar to that of other clinically used retinoids.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients who are diagnosed as probable Alzheimer' Disease according to NINCDS-ADRDA criteria
* Diagnosed by brain diagnostic imaging (CT, MRI) within six months before the consent and no occurrence of the event after that to suggest cerebral vascular disease
* Mild to Moderate Alzheimer's Disease of MMSE from 10 to 26
* Age from 55 to 80
* Treated for a minimum of 12 weeks with a stable dose of donepezil and willing to continue the same during the trial period
* For women Menopause ≥ 2 years
* For men contraceptive measures are required during the study and after 6 months
* In principle patients should be living at their home in the presence of a caregiver who is defined as a healthy person in contact with the patient for more than 10 hours a week, could provide required information of the behavior and activities of daily living, accompany all the clinical examination, and supervise the handling and administration of the drug throughout the study period.
* Patients who could take pills as a whole
* Patient, caregiver and patient surrogate are able and willing to comply with study visits and procedures per protocol, understand, sign, and date the written voluntary informed consent form

Exclusion Criteria:

* Any cause of dementia not due to Alzheimer's disease
* Past history of other central nervous condition or psychiatric disease
* Symptom of depression and drug addiction
* Impairment in the physical function by other factor than the Alzheimer's Disease
* Patients who are expected to move in to care facilities during the study period
* triglyceride > 400 mg/dL

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Alzheimer's Disease Assessment Scale (ADAS-JCog) | baseline, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Changes in Mini-Mental State Examination (MMSE) | baseline, 12 weeks, 24 weeks
Changes in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | baseline, 12 weeks, 24 weeks
Changes in Clinician Interview-Based Assessment of Change Plus Caregiver Information (CIBIC-Plus) | baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takami Miki, M.D., Principal Investigator — Department of Geriatrics and Neurology, Osaka City University Graduate School of Medicine
Locations (1):
- Osaka City University Hospital, Osaka, Japan

REFERENCES:
- [Background] Shudo K, Fukasawa H, Nakagomi M, Yamagata N. Towards retinoid therapy for Alzheimer's disease. Curr Alzheimer Res. 2009 Jun;6(3):302-11. doi: 10.2174/156720509788486581. PMID 19519313